CLINICAL TRIAL: NCT05736302
Title: Validating a New Machine-Learned Accelerometer Algorithm Using Doubly Labeled Water
Acronym: ValiDLW
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: University of Colorado, Denver (Other); University of Massachusetts, Amherst (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21.061; R01CA215318 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-08

CONDITIONS: Movement Disorders; Energy Metabolism
Keywords: Doubly labeled water (DLW); Total Daily Energy Expenditure (TDEE); Accelerometry
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine and Saliva- only retained until completion of data analysis, and then destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Individuals without movement limitations: Individuals who are not classified as impaired or functionally limited per results of physical function testing.
  Interventions: Other: Doubly-Labeled Water
- Individuals with impaired movement: Individuals who are classified as impaired, but not functionally limited per results of physical function testing.
  Interventions: Other: Doubly-Labeled Water
- Individuals with impaired movement who are functionally impaired: Individuals who are classified as impaired and functionally limited per results of physical function testing.
  Interventions: Other: Doubly-Labeled Water

INTERVENTIONS:
Other: Doubly-Labeled Water — All eligible participants will receive a dose of doubly-labeled water.

SUMMARY:
The purpose of this study is to validate previously developed physical function-clustered specific machine-learned accelerometer algorithms to estimate total daily energy expenditure (TDEE) in individuals with general movement and functional limitations.

DETAILED DESCRIPTION:
Current algorithms for examining accelerometer data were developed primarily using data from individuals without movement limitations or impairments. As such, the current available analytic algorithms are inadequate for use with individuals with limitations and impairments to estimate total daily energy expenditure (TDEE). The creation of a new algorithm that can accurately assess TDEE in individuals with movement limitations will be beneficial for future research examining physical activity interventions targeted to these individuals. This study will serve to validate a new algorithm that was developed specifically to analyze accelerometer data for individuals with movement limitations, and gauge the accuracy of the new algorithm's ability to accurately assess TDEE against one of the gold standards of TDEE measurement, the doubly labelled water technique.

Approximately 125 adults, 50 from Colorado, and 75 from Wisconsin, will participate in this study. Participants will complete three study visits. During the first visit, physical function will be assessed during a series of tests, and a dual-energy X-ray absorptiometry (DXA) scan will be performed to obtain information on body composition. During the second visit, the participant will complete a resting metabolic rate (RMR) examination, will consume a dose of doubly labeled water, and will provide urine and saliva samples. At the end of the second visit, participants will be given a set of accelerometers to wear for 8-10 days, and will be asked to complete a wear log for documentation. After 8-10 days have passed, during the final visit, participants will provide additional urine samples and return the accelerometers.

The hypothesis being tested is that physical function-clustered specific machine-learned accelerometer algorithms will produce more accurate and precise estimations of TDEE during free-living compared with healthy population derived accelerometer algorithms applied to diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* must be 18+ years of age
* be able to ambulate on own, unassisted, on a regular basis
* speak and read English
* must have access to a working smart phone and a computer with internet access

Exclusion Criteria:

* wheelchair reliant
* assistive walking device reliant (cannot walk for at least 50 feet without an assistive device)
* diagnosed uncontrolled hypertension (above 160/100 mgHg)
* diagnosed cognitive impairment or inability to follow study procedures such as Alzheimer's disease or dementia
* cannot take metabolic altering medications
* cannot be pregnant
* cannot be breastfeeding
* cannot use supplemental oxygen
* cannot completed required study activities for any reason
* cannot have a resting heart rate > 100 bpm or a resting blood pressure > 160 mgHg during Visit 1
* cannot weigh more than 450 lbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18+ years of age
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of accelerometer derived estimations of total daily energy expenditure (TDEE, kcals/day). | 8-10 days monitoring
  Accelerometer estimations will be derived by different algorithms available in the literature, as well as from a newly developed algorithm that distinguishes between those with and without movement limitations. Accelerometer estimations of TDEE will be compared to those values obtained by the criterion doubly-labeled water technique.
Precision of accelerometer derived estimations of total daily energy expenditure (TDEE, kcals/day). | 8-10 days monitoring
  Accelerometer estimations will be derived by different algorithms available in the literature, as well as from a newly developed algorithm that distinguishes between those with and without movement limitations. Accelerometer estimations of TDEE will be compared to those values obtained by the criterion doubly-labeled water technique.
Total Daily Energy Expenditure (TDEE) (via DLW) | pre-dose; 4 hours and 5 hours post-dose, and 8-10 days post-dose
  Total daily energy expenditure (TDEE) over the 8-10 day period as measured by the difference in presence of isotopes in the samples at Visit 3. The 18-O and deuterium exit the body through slightly different mechanisms, so when we examine the difference in levels present at the end of the 8-10 day period between Visit 2 and Visit 3, we can estimate carbon dioxide (CO2) production and hence, energy expenditure. The samples taken at Visit 2 provide the baseline information required to analyze the samples taken at Visit 3 and calculate TDEE.

SECONDARY OUTCOMES:
Resting Metabolic Rate (kcals/day) | pre-dose
  Basal metabolic rate as determined by fasting RMR test, conducted via Parvomedics TrueOne 2400 Metabolic system. Results include the approximate number of calories an individual would expend if they spent the day in a resting state.
Fat free body mass (g) | 7-14 days before dose
  Dual x-ray absorptiometry (DEXA) measurement of body composition, conducted via a Hologic Horizon W system. Results include the amount of fat, bone mineral density, and fat free mass, measured in grams. The fat free mass measurement is used to calculate the dose of doubly labeled water for the participant.
Modified Physical Performance Test (MPPT) | 7-14 days before dose
  The modified physical performance test consists of 9 subtests that are used to assess level of physical function. Total scores range from 0-36. Not frail = 32-36, Mildly frail = 25-31, Moderately frail = 17-24, and less than 17= low function.
Maximum hand grip strength | 7-14 days before dose
  Hand grip is measured via a hand grip dynamometer manufactured by Lafayette Instruments, and is equivalent to the Jamar hand grip dynamometer. The results are measured in lbs, and can range from 0 lbs to 250 lbs. Cut offs for normal hand grip strength vary significantly dependent upon age, sex, country of origin, and BMI. Lower hand grip strength is associated with lower physical function.
Gait speed | 7-14 days before dose
  Gait speed is measured via the 10 meter walk test, with three repetitions of the test at a normal walking speed, and three repetitions of the test at a fast walking speed. A number of different published cut-offs exist for this test, but a cut-off of 1.0 m/sec is recognized as being an indicator of lower physical function. Individuals who ambulate slower than 1.0 m/sec are at risk of not being able to function in the community.
Temporospatial gait analysis | 7-14 days before dose
  Analysis of gait to determine whether anomalies are present via the GAITrite system. Over 50 variables are taken into account in the analysis. These results are compared to standardized norms (sex and age based), and elements of the analysis that are abnormal compared to those norms are indicated in the system output.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Strath, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided
Following completion of the study, all accrued data will be handled and collated in a manner consistent to allow for dissemination of generated data sets to qualified researchers in the scientific community for further analyses and study.